CLINICAL TRIAL: NCT04088422
Title: Prospective, Observational Study on Cell Free DNA Genotyping as a Tool to Inform Mature B-cell Lymphoma Management
Brief Title: Cell Free DNA in Mature B-cell Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Other Study IDs: cfDNA
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Mature B-Cell Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- B-cell lymphoma
  Interventions: Procedure: peripheral blood collection

INTERVENTIONS:
Procedure: peripheral blood collection — peripheral blood collection at treatment start, interm PET/CT, end of treatment PET/CT, one-year and two-year follow-up and or progression or relapse

SUMMARY:
The purpose of this study is to assess whether plasma cell free DNA is an accurate tool that can early and dynamically inform on treatment outcome and an accessible source of tumor DNA to track tumor clonal evolution.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of mature B-cell tumor according to WHO 2008 criteria
* 18 years or older

Exclusion Criteria:

* Chemotherapy before
* Other tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of mature B-cell tumor according to WHO 2008 criteria without any previous treatment in Ruijin Hospital would be included.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2-year

SECONDARY OUTCOMES:
overall survival | 2-year
Complete Response rate | 6 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD，PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China